CLINICAL TRIAL: NCT02497807
Title: fMRI Study on Iron Deficiency in the Pathological Mechanism of Tourette Syndrome
Brief Title: The Pathophysiology of Tourette Syndrome: a Multimodal Study
Acronym: PTS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian Hua Feng, professor of medicine, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: SAHZJU_CCBD_TouretteS
Record Dates: First submitted 2014-05-13; First posted 2015-07-15 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Tourette Syndrome
Keywords: Tourette syndrome; Iron deficiency
MeSH Terms: conditions — Tourette Syndrome; Iron Deficiencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: None Retained — no biospecimens are to be retained
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to characterize the functional and anatomical connectivity changes in Tourette syndrome and its relation with iron deficiency.

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a childhood-onset chronic neuropsychiatric disorder with an increasing prevalence (range 0.05-3%).The investigators previous study showed that lower serum ferritin and iron levels in children with Tourette syndrome than in healthy children. The exact mechanism explaining how iron deficiency contributes to the pathophysiology of TS is unclear.One question is whether or not peripheral iron deficiency in children with Tourette syndrome can inflence the brain extrapyramid structure and resting state brain function？Another question is how well peripheral iron indices correlate with central iron content？ The third question is for TS children with peripheral iron deficiency, oral iron supplement (5mg/Kg/d) at least 8 weeks, the peripheral iron indicies return to normal levels, how the brain iron contents and the relative structure and brain function change?, To test the above-metioned hypothesis, functional magnetic resonance imaging (fMRI) , diffusion tensor imaging (DTI) and susceptibility weighted imaging (SWI) are applied to investigate the volume change of extrapyramid structure such as caudate nucleus and putamen, resting-state brain function and brain iron content before and after oral iron supplementation in TS children with peripheral iron deficiency, TS children with peripheral normal iron levels and normal healthy controls. The investigators hope to confirm that iron deficiency may play a causal role in the dopamine metabolism and it helps to further explore the pathophysiology of Tourette syndrome and also would contribute to significant advance in the therapeutic option for TS children with peripheral iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years old
* Characterized by vocal tic and muscle twitch
* No positive signs was found through neurological examination, no significant psychomotor retardation,

Exclusion Criteria:

* Hepatolenticular degeneration
* Rheumatic chorea
* Myoclonic epilepsy
* History of mental disease or brain trauma

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients were recruited from outpatients or inpatients with Tourette syndrome.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-11 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Amplitude of low frequency fluctuation of BOLD signal in Tourette syndrome and its relation with iron deficiency | two years
  Amplitude of low frequency fluctuation of BOLD signal has proven to be a promising way to detect disease-related local brain activity.This study investigate ALFF in Tourette syndrome and provides insights into the pathological mechanism of Tourette syndrome

SECONDARY OUTCOMES:
Brain iron levels in Tourette syndrome | two years

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Feng, Doctor, Principal Investigator — Second affiliated hospital,zhejiang University,school of medicine,; Jianhua Feng, Doctor, Principal Investigator — Secon Affiliated Hospital,Zhejiang University,School of Medicine
Locations (1):
- Second Affiliated Hospital,Zhejiang University,School of Medicine, Hangzhou, Zhejiang, China